CLINICAL TRIAL: NCT06245486
Title: Study on the Efficacy of Crispact® (Probiotic Containing Lactobacillus Crispatus M247) in the Sterilization of HPV-HR and in the Reconstitution of the Normal Vaginal Microbiota
Brief Title: Probiotc Lactobacillus Crispatus-M247 (Crispact®) Supplementation in the Sterilization of High-risk Human Papilloma (HPV-HR) Viruses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 774/18.10.2021
Record Dates: First submitted 2024-01-20; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Probiotic Crispact® (20 Bld CFU/Stick of Lactobacillus crispatus M247)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotic Young Group (Women aged 18-29 years) (Experimental): Participants in this group will take probiotic Crispact® (20 Bld CFU/Stick of Lactobacillus crispatus M247) as 1 oral sachet per day for four months and 1 sachet in vaginal lavage for the first 10 days of treatment.
  Interventions: Dietary Supplement: Crispact®
- Control Young Group (Women aged 18-29 years) (Active Comparator): Participants in this group will take Placebo as 1 oral sachet per day for four months and 1 sachet in vaginal lavage for the first 10 days of treatment.
  Interventions: Dietary Supplement: Placebo
- Probiotic Lady Group (Women aged 30-64 years) (Experimental): Participants in this group will take probiotic Crispact® (20 Bld CFU/Stick of Lactobacillus crispatus M247) as 1 sachet oral per day for four months and 1 sachet in vaginal lavage for the first 10 days of treatment.
  Interventions: Dietary Supplement: Crispact®
- Control Lady Group (Women aged 18-29 years) (Active Comparator): Participants in this group will take Placebo as 1 oral sachet per day for four months and 1 sachet in vaginal lavage for the first 10 days of treatment.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Crispact® — Contains 20 Bld CFU/Stick of probiotic Lactobacillus crispatus M247
  Arms: Probiotic Lady Group (Women aged 30-64 years); Probiotic Young Group (Women aged 18-29 years)
Dietary Supplement: Placebo — Placebo
  Arms: Control Lady Group (Women aged 18-29 years); Control Young Group (Women aged 18-29 years)

SUMMARY:
There is growing scientific interest in probiotic supplementation as a possible therapy for clearing the human papillomavirus (HPV) infection and reducing the risk of developement of cervical cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, longitudinal, prospective, parallel-group, single-blind study aimed to investigate the efficacy of probiotic Crispact® (which contains: 20 Bld CFU/Stick of Lactobacillus crispatus M247) in clearance of human papillomavirus (HPV) infection in healthy female who tested positive for human papillomavirus (HPV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Women able to understand and agree to participation in the study and be able to provide written informed consent to the trial.
* Women aged 25-29 years who perform screening pap smears with the result: Low- grade squamous intraepithelial lesion (LSIL) or Atypical Squamous Cells of Undetermined Significanc (ASCUS) (for which, as per the recommendation of the Italian Society of Colposcopy and Cervico-Vaginal Pathology (SICPCV)/Italian Group of Cervical Cancer. Screening (GISCI), no treatment is indicated but only follow-up with Human papillomavirus (HPV) test at 12 months.
* Women aged 18-64 who independently perform a positive High risk sub-types of HPV (HR-HPV) test outside of screening even in the presence of a negative cytology (for whom, as per the recommendation of the SICPCV, no treatment is indicated but only follow-up with HPV test at 12 months).
* Women aged 30-64 years HPV HR positive with negative cytology or with positive cytology for ASCUS or LSIL but negative colposcopy (absence of colposcopic lesion or positive colposcopy but subsequent negative biopsy) who do not require treatment (therefore as per the recommendation of the SICPCV go to follow-up with HPV testing at 12 months).

Exclusion Criteria:

* Women who have been vaccinated for HPV.
* Patients who have undergone cervical treatments for preneoplastic pathology.
* Patients with High-Grade Squamous Intraepithelial Lesion (HSIL) cytological result who on histological examination after biopsy need treatment according to the SICPCV 2019 recommendations.
* Hypersensitivity to one or more components of the product.
* Patients being treated with antibiotic, immunomodulatory and immunosuppressive therapies.
* Patients with immune system or neoplastic pathologies being treated with chemotherapy
* Patients who are pregnant, breastfeeding, or planning to become pregnant in the next 6 months.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is only applicable in women
Enrollment: 150 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Human papillomavirus (HPV) clearance | After 4-months
  Testing negative for HPV
Changes in vaginal bacterial quantity (population) that colonize, called Community State Type (CST) | After 4-months
  Changes in vaginal microbiota

IPD SHARING:
Plan to Share IPD: No